CLINICAL TRIAL: NCT00858234
Title: A Multicenter, Open-Label, Phase I Study of MK-0683 in Combination With Bortezomib in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Phase I Study of MK-0683 in Combination With Bortezomib in Participants With Multiple Myeloma (MK-0683-098)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0683-098; MK-0683-098 (Other: Merck)
Record Dates: First submitted 2009-03-04; First posted 2009-03-09 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat + Bortezomib (Experimental): Participants undergo up to 3 successive 21-day treatment cycles. During Cycle 1, participants receive vorinostat (400 mg once daily [QD] on Days 1 through 14) + bortezomib (1.3 mg/m^2 intravenous [IV] on Days 1, 4, 8, and 11). If that dose is not well tolerated, during Cycle 2 participants receive vorinostat (400 mg QD on Days 1 through 14) + bortezomib (1.0 mg/m^2 IV on Days 1, 4, 8, and 11). If that dose is not well tolerated, during Cycle 3 participants receive vorinostat (300 mg QD on Days 1 through 14) + bortezomib (1.0 mg/m^2 IV on Days 1, 4, 8, and 11).
  Interventions: Drug: Vorinostat; Drug: Bortezomib

INTERVENTIONS:
Drug: Vorinostat — Vorinostat (MK-0683) three or four 100 mg capsules taken by mouth with food.
  Other Names: MK-0683; ZOLINZA™
Drug: Bortezomib — Bortezomib (1.0 or 1.3 mg/m^2) intravenous infusion.
  Other Names: VELCADE®

SUMMARY:
The primary purpose of this clinical study is to determine the recommended clinical doses of vorinostat (MK-0683) and bortezomib administered in combination to participants with relapsed and/or refractory multiple myeloma (MM). It was hypothesized that administration of vorinostat in combination with bortezomib is sufficiently safe and tolerated well enough to permit further study in participants with relapsed and/or refractory MM. Study results are based on data collected up to the data cut-off date of 20-March-2011.

ELIGIBILITY:
Inclusion Criteria:

* is ≥20 years of age.
* has an established diagnosis of MM based on the myeloma diagnostic criteria
* has received at least 1 but not more than 3 prior anti-myeloma regimens and has progressive disease after the most recent treatment regimen
* has adequate organ function

Exclusion Criteria:

* has had a prior allogeneic bone marrow transplant or plans to undergo any type of bone marrow transplantation during the study
* has known hypersensitivity to any components of vorinostat or bortezomib
* has active hepatitis B or C, plasma cell leukemia, or is human immunodeficiency virus (HIV) positive
* has had prior treatment with vorinostat or histone deacetylase (HDAC) inhibitors

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-02-13 (Actual); Primary Completion 2010-06-11 (Actual); Study Completion 2012-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ogawa Y, Ogura M, Tobinai K, Ando K, Suzuki T, Watanabe T, Ohmachi K, Uchida T, Hanson ME, Tanaka Y, Koh Y, Shimamoto T, Hotta T. A phase I study of vorinostat combined with bortezomib in Japanese patients with relapsed or refractory multiple myeloma. Int J Hematol. 2016 Jan;103(1):25-33. doi: 10.1007/s12185-015-1897-7. Epub 2015 Nov 30. PMID 26619834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants with relapsed and/or refractory multiple myeloma (MM) were enrolled at study sites in Japan.
Groups:
- Vorinostat + Bortezomib: Participants undergo ≤3 successive 21-day treatment cycles. During Cycle 1, participants receive vorinostat (400 mg QD on Days 1 through 14) + bortezomib (1.3 mg/m^2 IV on Days 1, 4, 8, and 11). If that dose is not well tolerated, during Cycle 2 participants receive vorinostat (400 mg QD on Days 1 through 14) + bortezomib (1.0 mg/m^2 IV on Days 1, 4, 8, and 11). If that dose is not well tolerated, during Cycle 3 participants receive vorinostat (300 mg QD on Days 1 through 14) + bortezomib (1.0 mg/m^2 IV on Days 1, 4, 8, and 11).
Period: Overall Study
Arm/Group | Vorinostat + Bortezomib
Started | 9
Completed | 0
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Progressive disease | 2
Not completed — Status unknown | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) During Cycle 1
Description: The number of participants with ≥1 DLT during Cycle 1 is reported. A DLT is defined as an event considered by the investigator to be related to study treatment, and either: 1) a Grade 3 or 4 non-hematologic event (except for manageable toxicity by supportive care or non-prohibited therapies, or a transient increase in alanine aminotransferase [ALT]/aspartate aminotransferase [AST]); or 2) a Grade 4 hematologic toxicity except neutropenia or hemoglobin decreased (neutropenia was a DLT if it was Grade 3-4 with fever ≥38.5°C; Grade 3-4 with an infection requiring antibiotic/antifungal therapy; or Grade 4 and lasting ≥5 days).
Time Frame: Up to 21 days
Population: All treated participants who were not refractory to bortezomib and met all inclusion criteria are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 6
Participants | 1

2. Other Pre Specified Outcome: Number of Participants With an Adverse Event (AE)
Description: The number of participants with ≥1 AE is reported. An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product(s), whether or not considered related to the use of the product(s).
Time Frame: Up to 346 days (up to 30 days after the final dose of study treatment)
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 9
Participants | 9

3. Other Pre Specified Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours Postdose (AUC0-24hr) of Vorinostat Administered With Bortezomib on Days 1 and 11
Description: The AUC0-24hr of vorinostat in plasma on Days 1 and 11 is reported in participants who also received bortezomib.
Time Frame: Predose and 0.8, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose on Days 1 and 11
Population: Participants with data available are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 9
µM*hr
  Day 1 | 5.41 [4.33 to 6.77]
  Day 11: number analyzed (Participants) | 7
  Day 11 | 5.84 [4.48 to 7.61]
Statistical Analysis 1: Comparison: Vorinostat + Bortezomib; Test type: Other — Accumulation Ratio (Day 11 AUC0-24hr/Day 1 AUC0-24hr); Accumulation ratio = 1.08, 90% CI 2-sided [0.80 to 1.45] — Back-transformed least squares mean difference and 90% confidence interval from mixed effects model performed on natural log-transformed values

ADVERSE EVENTS:
Time Frame: Up to 346 days (up to 30 days after the final dose of study treatment)
Description: All treated participants are included.
Arm/Group | Vorinostat + Bortezomib
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat + Bortezomib (N=9)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat + Bortezomib (N=9)
Anaemia (Blood and lymphatic system disorders) | 3 (8)
Leukopenia (Blood and lymphatic system disorders) | 9 (98)
Lymphopenia (Blood and lymphatic system disorders) | 6 (32)
Neutropenia (Blood and lymphatic system disorders) | 9 (99)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (189)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (16)
Diarrhoea (Gastrointestinal disorders) | 9 (44)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (31)
Stomatitis (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 7 (19)
Fatigue (General disorders) | 5 (18)
Injection site reaction (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (9)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood albumin decreased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 2 (9)
Blood glucose increased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2)
Blood potassium increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (4)
Electrocardiogram ST-T segment depression (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 8 (24)
Dehydration (Metabolism and nutrition disorders) | 2 (4)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (20)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (24)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 1 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.